CLINICAL TRIAL: NCT01887587
Title: Phase I Study Of Vincristine, Doxorubicin, And Dexamethasone (VXD) Plus Ixazomib In Adults With Relapsed Or Refractory Acute Lymphoblastic Leukemia/Lymphoma, Lymphoblastic Lymphoma Or Mixed Phenotype Acute Leukemia
Brief Title: Vincristine, Doxorubicin, And Dexamethasone + Ixazomib in Acute Lymphoblastic Leukemia (ALL), Lymphoblastic Lymphoma Or Mixed Phenotype Acute Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: SAE- risk of overall protocol treatment outweighs benefits
Sponsor: Ehab L Atallah (Other)
Responsible Party: Sponsor-Investigator, Ehab L Atallah, Associate Professor, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00020384
Record Dates: First submitted 2013-06-05; First posted 2013-06-27 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2019-12

CONDITIONS: Relapsed or Refractory Acute Lymphoblastic Leukemia; Relapsed or Refractory Lymphoblastic Lymphoma; Mixed Phenotype Acute Leukemia
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute | interventions — ixazomib; Vincristine; Doxorubicin; liposomal doxorubicin; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- (modified VXLD) plus MLN9708 (Experimental): Vincristine-1.5 mg/m2 to a max dose of 2 mg IV on days 1, 8, 15 and 22
  Dexamethasone- 10 mg/m2 orally or IV on days 1-14
  Doxorubicin- 60 mg/m2 on day 1 by IV bolus.
  MLN9708 (Ixazomib)- 2.3 mg orally on days 1, 8 and 15. Escalations will be to 3mg or 4 mg, respectively, on days 1, 8 and 15 based on the dosing schema.
  For patients without central nervous system (CNS) involvement:
  * Cytarabine 100 mg administered intrathecally on day 1 (cytarabine dose should be reduced to 50 mg if given through a central ommaya reservoir)
  * Methotrexate 12 mg administered intrathecally on day 8
  For patients with CNS involvement:
  -Cytarabine 100 mg administered intrathecally on day 1 (+/-1 day) (cytarabine dose should be reduced to 50 mg if given through a central ommaya reservoir) Triple intrathecal chemotherapy with cytarabine 30 mg, methotrexate 15 mg and hydrocortisone 15 mg on (Day 1, 8, 15 and 22 (+/-1 day)).
  Interventions: Drug: MLN9708; Drug: Vincristine; Drug: Doxorubicin; Drug: Dexamethasone

INTERVENTIONS:
Drug: MLN9708
  Other Names: Ixazomib
Drug: Vincristine
  Other Names: Oncovin
Drug: Doxorubicin
  Other Names: Doxil; hydroxydaunorubicin
Drug: Dexamethasone
  Other Names: Decadron; Dexasone; Solurex; Baycadron

SUMMARY:
This is a phase I study of vincristine, doxorubicin and dexamethasone (modified VXD) plus MLN9708 in adults with relapsed or refractory acute lymphoblastic leukemia/lymphoma, lymphoblastic lymphoma or mixed phenotype acute leukemia.

DETAILED DESCRIPTION:
In this phase I study, escalating doses of MLN9708 will be combined with a fixed dose modified VXD regimen. The study drug, MLN9708, will be administered on day 1, 8, and 15. If the patient experiences a dose limiting toxicity (DLT) the dose of MLN9708 maybe reduced to the next dose level on day 8 or day 15 in that patient. DLT would be any grade 3 or more toxicity which is thought to be probably or definitely related to MLN9708. Three patients will be treated per dose level unless DLT is observed. The starting dose of MLN9708 will be 2.3 mg orally on days 1, 8 and 15. If toxicity is seen at this level then dose may be reduced to 1.5 mg (dose level -1) . If no DLT is seen in the first 3 patients, the dose will be increased to 3 mg and then to 4 mg orally on days 1, 8 and 15 in a classic 3 +3 phase I design. We will not attempt to increase the dose beyond 4 mg orally which, if achieved with acceptable toxicity, would be accepted as the recommended phase 2 dose (RP2D). 0 of 3 DLTs would allow escalation to the next dose level. 1 of 3 DLTs will require expanding to six patients; 1 of 6 DLTs will allow escalation again. 2 DLTs will require dose de-escalation. The maximum tolerated dose (MTD) will be the highest dose administered at which no more than 1 DLT was observed. All patients will be evaluated for hematopoetic stem cell transplantation. If patients achieve complete response (CR) and are eligible for hematopoietic stem cell transplantation (HSCT), they will proceed to HSCT. If they are not eligible, no donor is identified or if HSCT will be delayed, and the patient has achieved benefit, then treatment maybe repeated at the discretion of the investigator. A total of 9-18 patients will be enrolled on the study. The study duration would be about 2 years.

ELIGIBILITY:
Each patient must meet all of the following inclusion criteria to be enrolled in the study:

Inclusion

* Male or female patients 18 years or older
* Have relapsed B or T-precursor acute lymphocytic leukemia/lymphoma, lymphoblastic lymphoma or mixed phenotype acute leukemia with increased bone marrow or peripheral blood blasts by morphology with or without CNS involvement
* Prior therapy: At least two prior treatment attempts to induce remission with no limit on the number of prior treatment regimens.
* Patients are eligible after allogeneic stem cell transplantation
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must meet the following clinical laboratory criteria:

  * Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
  * Calculated creatinine clearance ≥ 30 mL/min
  * Absolute neutrophil count (ANC) > 1,000/cmm and platelets > 75,000/cmm unless the cytopenias are secondary to disease
* Life expectancy reasonably adequate for evaluating the treatment effect
* Patients must be at least 2 weeks from major surgery, radiation therapy, participation in other investigational trials and have recovered from clinically significant toxicities of these prior treatments
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.).

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Patients who are Ph+ ALL who are naive to therapy with an approved tyrosine kinase inhibitor.
* Prior exposure to ≥350 mg/m2 of anthracycline (in doxorubicin equivalent dosing), or left ventricular fractional shortening less than 50%.
* Failure to have fully recovered (ie, ≤ Grade 2 toxicity) from the effects of prior chemotherapy regardless of the interval since last treatment.
* Major surgery within 14 days before enrollment.
* Chemotherapy in the last 14 days. (Steroids or Intrathecal chemotherapy will be allowed).
* Systemic treatment, within 7 days before study enrollment, with strong inhibitors of cytochrome P450 1A2 (CYP1A2) (e.g., fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of cytochrome P4503A (CYP3A) (e.g., clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, or psychiatric illness/social situations that would limit compliance with study requirements. Patients receiving intravenous antibiotics for infections that are under control may be included in this study.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or GI procedure that could interfere with the oral absorption or tolerance of treatment.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Patient has ≥ Grade 2 peripheral neuropathy.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Female patients who are breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-06; Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ehab L Atallah, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- (Modified VXLD) Plus MLN9708: Vincristine-1.5 mg/m2 to a max dose of 2 mg IV on days 1, 8, 15 and 22
  Dexamethasone- 10 mg/m2 orally or IV on days 1-14
  Doxorubicin- 60 mg/m2 on day 1 by IV bolus.
  For patients without central nervous system (CNS) involvement:
  * Cytarabine 100 mg will be administered intrathecally on day 1 (+/-1 day) (cytarabine dose should be reduced to 50 mg if given through a central ommaya reservoir)
  * Methotrexate 12 mg will be administered intrathecally on day 8 (+/-1 day)
  For patients with CNS involvement:
  -Cytarabine 100 mg will be administered intrathecally on day 1 (+/-1 day) (cytarabine dose should be reduced to 50 mg if given through a central ommaya reservoir) Triple intrathecal chemotherapy with cytarabine 30 mg, methotrexate 15 mg and hydrocortisone 15 mg on (Day 1, 8, 15 and 22 (+/-1 day)).
Period: Overall Study
Arm/Group | (Modified VXLD) Plus MLN9708
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- (Modified VXLD) Plus MLN9708: Vincristine-1.5 mg/m2 to a max dose of 2 mg IV on days 1, 8, 15 and 22
  Dexamethasone- 10 mg/m2 orally or IV on days 1-14
  Doxorubicin- 60 mg/m2 on day 1 by IV bolus.
  For patients without CNS involvement:
  * Cytarabine 100 mg will be administered intrathecally on day 1 (+/-1 day) (cytarabine dose should be reduced to 50 mg if given through a central ommaya reservoir)
  * Methotrexate 12 mg will be administered intrathecally on day 8 (+/-1 day)
  For patients with CNS involvement:
  -Cytarabine 100 mg will be administered intrathecally on day 1 (+/-1 day) (cytarabine dose should be reduced to 50 mg if given through a central ommaya reservoir) Triple intrathecal chemotherapy with cytarabine 30 mg, methotrexate 15 mg and hydrocortisone 15 mg on (Day 1, 8, 15 and 22 (+/-1 day)).
  MLN9708
  Vincristine
  Doxorubicin
  Dexamethasone
Arm/Group | (Modified VXLD) Plus MLN9708
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 49 [25 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events.
Description: Safety, tolerability will be assessed by counting the number of participants experiencing adverse events at 8 weeks post treatment.
Time Frame: Baseline to 30 days post treatment; approximately 8 weeks
Population: At dose level one, 3 patients who were enrolled. The protocol was amended to remove PEGaspargase from the regimen. Two additional patients were enrolled on dose level one.
Measure: Number; unit: participants
Arm/Group | (Modified VXLD) Plus MLN9708
Number analyzed (Participants) | 5
participants | 5

2. Primary Outcome: Optimal Dose of MLN9708
Description: This measure will be the maximum tolerated dose (MTD) at which no more than 1 Dose Limiting Toxicity (DLT) is observed. The starting dose of MLN9708 will be 2.3 mg orally on days 1, 8 and 15. If no DLT is seen in the first 3 patients, the dose will be increased to 3 mg and then to 4 mg orally on days 1, 8 and 15 in a classic 3 +3 phase I design. We will not attempt to increase the dose beyond 4 mg orally which, if achieved with acceptable toxicity, would be accepted as the recommended phase 2 dose (RP2D). 0 of 3 DLTs would allow escalation to the next dose level. 1 of 3 DLTs will require expanding to six patients; 1 of 6 DLTs will allow escalation again. 2 DLTs will require dose de-escalation.
Time Frame: 8 Weeks
Population: All five subjects received the same 2.3 mg oral dose of MLN9708.
Measure: Number; unit: mg
Groups:
- Modified VXLD Plus MLN9708: Vincristine -1.5 mg/m2 to a max dose of 2 mg IV on days 1, 8, 15 and 22
  Dexamethasone - 10 mg/m2 orally or IV on days 1-14
  Doxorubicin - 60 mg/m2 on day 1 by IV bolus.
  MLN9708 (Ixazomib)- 2.3 mg orally on days 1, 8 and 15. Subsequent escalations will be to 3mg or 4 mg, respectively, on days 1, 8 and 15 based on the dosing schema.
  For patients without CNS involvement:
  * Cytarabine 100 mg will be administered intrathecally on day 1 (+/-1 day) (cytarabine dose should be reduced to 50 mg if given through a central ommaya reservoir)
  * Methotrexate 12 mg will be administered intrathecally on day 8 (+/-1 day)
  For patients with CNS involvement:
  -Cytarabine 100 mg will be administered intrathecally on day 1 (+/-1 day) (cytarabine dose should be reduced to 50 mg if given through a central ommaya reservoir) Triple intrathecal chemotherapy with cytarabine 30 mg, methotrexate 15 mg and hydrocortisone 15 mg on (Day 1, 8, 15 and 22 (+/-1 day).
Arm/Group | Modified VXLD Plus MLN9708
Number analyzed (Participants) | 5
mg | 2.3

ADVERSE EVENTS:
Time Frame: 8 weeks following last dose.
Arm/Group | (Modified VXLD) Plus MLN9708
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (Modified VXLD) Plus MLN9708 (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Sepsis (Infections and infestations) | 3
Methemoglobinemia (Investigations) | 1
Sinus tachycardia (Cardiac disorders) | 1
Lactic acidosis (Hepatobiliary disorders) | 1
Increased blood bilirubin (Hepatobiliary disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-06-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT01887587/Prot_SAP_000.pdf
  • Informed Consent Form (2015-08-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT01887587/ICF_001.pdf